CLINICAL TRIAL: NCT03591146
Title: A Phase I/II, Randomized, Double-blind, Comparator-controlled, Dose-escalation Study to Evaluate the Safety, Pharmacokinetics, and Efficacy of TLC590 for Postsurgical Pain Management Following Inguinal Hernia Repair
Brief Title: Phase I/II Dose-escalation Study to Evaluate Safety, PK and Efficacy of TLC590 for Postsurgical Pain Management
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Taiwan Liposome Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: TLC590A1001
Record Dates: First submitted 2018-06-25; First posted 2018-07-19 (Actual); Results first posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-06

CONDITIONS: Inguinal Hernia
Keywords: Postsurgical Pain Management
MeSH Terms: conditions — Hernia, Inguinal | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: Subjects will be enrolled to each cohort in a 3:1 ratio. Each cohort will comprise subjects receiving a dose of TLC590 and active comparator drug (Naropin® 150 mg) in accordance with the randomization schedule and dose-escalation scheme.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: To maintain objectiveness, the study drug will be managed and administered by an independent unblinded team. Subjects, investigators, and all other site staff who directly interact with subjects, evaluate safety and efficacy, and collect subject data, will remain blinded and must not communicate or discuss any study information with the unblinded team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- TLC590 190mg (Experimental): TLC590 (Ropivacaine Liposome Injectable Suspension) is a sustained-release liposome formulation of ropivacaine, white aqueous suspension with ropivacaine concentration at approximately 19 mg/mL.
  Interventions: Drug: TLC590
- TLC590 380mg (Experimental): TLC590 (Ropivacaine Liposome Injectable Suspension) is a sustained-release liposome formulation of ropivacaine, white aqueous suspension with ropivacaine concentration at approximately 19 mg/mL.
  Interventions: Drug: TLC590
- TLC590 570mg (Experimental): TLC590 (Ropivacaine Liposome Injectable Suspension) is a sustained-release liposome formulation of ropivacaine, white aqueous suspension with ropivacaine concentration at approximately 19 mg/mL.
  Interventions: Drug: TLC590
- TLC590 475mg (Experimental): TLC590 (Ropivacaine Liposome Injectable Suspension) is a sustained-release liposome formulation of ropivacaine, white aqueous suspension with ropivacaine concentration at approximately 19 mg/mL.
  Interventions: Drug: TLC590
- Naropin 150mg (Active Comparator): Naropin injection contains ropivacaine hydrochloride (HCl). Strength: 150mg/ 30mL (5 mg/mL) Size: 30mL fill, in a 30mL single dose vial
  Interventions: Drug: Naropin

INTERVENTIONS:
Drug: TLC590 — TLC590 lyophilized cake will be reconstituted with the TLC590 reconstitution solution to form the TLC590 ropivacaine liposome injectable suspension
  Other Names: TLC590 (Ropivacaine Liposome Injectable Suspension)
  Arms: TLC590 190mg; TLC590 380mg; TLC590 475mg; TLC590 570mg
Drug: Naropin — Local infiltration of Naropin to produce anesthesia for surgery and analgesia in postoperative pain management. Naropin 150mg [0.5%, 5mg/mL] x 30mL
  Other Names: Naropin, 0.5% Injectable Solution
  Arms: Naropin 150mg

SUMMARY:
Phase I/II, randomized, double-blind, comparator-controlled, dose-escalation study to assess the safety, PK, and efficacy of single postsurgical application of TLC590 compared with Naropin®

DETAILED DESCRIPTION:
A Phase I/II, randomized, double-blind, comparator-controlled, dose-escalation study to assess the safety, PK, and efficacy of single postsurgical application of TLC590 compared with Naropin® via a single infiltrative local administration in adult subjects following inguinal hernia repair surgery.

Approximately 64 evaluable subjects across 4 cohorts. Dose escalation of a single postsurgical administration of TLC590 or Naropin® will be performed. Dose escalation will be determined by review of treatment-related adverse events and all serious adverse events (AEs) by a safety monitoring committee.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent.
2. Male or female between 18 and 65 years of age.
3. Scheduled to undergo a primary, unilateral Lichtenstein inguinal hernia repair with mesh, and be able to use the anesthesia regimen.
4. American society of anesthesiologists (ASA) Physical Status Classification of 1 or 2.
5. Female subjects are eligible only if: not pregnant; not lactating; not planning to become pregnant during the study; commits to the use of an acceptable form of birth control.
6. Male subjects must be sterile or commit to the use of a reliable method of birth control for the duration of the study until at least 1 week after the administration of blinded study medication.
7. Body mass index ≤ 35 kg/m2.

Exclusion Criteria:

1. Clinically significant abnormal clinical laboratory test value.
2. Evidence of a clinically significant 12-lead ECG.
3. History or evidence of orthostatic hypotension, syncope or other syncopal attacks.
4. History or clinical manifestations of significant renal, hepatic, gastrointestinal, cardiovascular, metabolic, neurologic, psychiatric, or other condition.
5. History of seizures or are currently taking anticonvulsants.
6. History of hypersensitivity to ropivacaine, any other amide-type local anesthetic, propofol, hydromorphone or oxycodone (or other opioids).
7. Persistent or recurrent nausea and/or vomiting due to other etiologies, including, but not limited to gastric outlet obstruction, hypercalcemia, or active peptic ulcer.
8. History of severe or refractory post-operative nausea or vomiting deemed clinically significant.
9. Concurrent painful condition that may require analgesic treatment during the study period.
10. Have been receiving or have received chronic opioid therapy.
11. Use of any of the following medications within 5 half-lives or as specified prior to the study surgical procedure:

    Anti-platelet agents such as aspirin therapy within 7 days; clopidogrel within 5 days; Anticoagulants such as warfarin within 5 days; dabigatran etexilate mesylate within 2 days; factor Xa inhibitor within 24 hours; Class III antiarrhythmic drugs (e.g., amiodarone); Strong CYP1A2 inhibitors, such as cimetidine, ciprofloxacin, enoxacin, and fluvoxamine; CYP1A2 substrates, such as theophylline or imipramine; Strong CYP3A4 inhibitors such as voriconazole, erythromycin, ketoconazole, or ritonavir; CYP3A4 substrates, such as atazanavir, darunavir, indinavir, lopinavir, nelfinavir, ritonavir, saquinavir, or tipranavir; Corticosteroids, either systemically, inhaled, intranasally, orally, or by intra-articular injection within 14 days before the study surgical procedure (topical corticosteroid is allowed); Non-steroidal anti-inflammatory drugs (NSAIDs) within 14 days prior to the study surgical procedure; Any investigational product within 30 days prior to administration of blinded study medication.
12. History of alcohol abuse or prescription and/or illicit drug abuse within 2 years.
13. Current report of alcohol abuse within 6 months.
14. Positive results on the urine drug screen or alcohol breath test indicative of illicit drug or alcohol abuse.
15. History of human immunodeficiency virus (HIV), hepatitis C, or hepatitis B.
16. Have had an inguinal hernia repair in the last 3 months before the study surgical procedure or presents with bilateral or recurrent inguinal hernia, other hernia presentations, or hernias with a large scrotal component that would be difficult to reduce surgically.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2019-01-05 (Actual); Study Completion 2019-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl Brown, PhD, Study Director — Taiwan Liposome Company
Locations (1):
- JBR Clinical Research, Draper, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Naropin 150mg: Naropin injection contains ropivacaine HCl. Strength: 150mg/ 30mL (5 mg/mL) Size: 30mL fill, in a 30mL single dose vial
  Naropin: Local infiltration of Naropin to produce anesthesia for surgery and analgesia in postoperative pain management. Naropin 150mg [0.5%, 5mg/mL] x 30mL
Period: TLC590 190mg and Naropin 150mg
Arm/Group | TLC590 190mg | TLC590 380mg | TLC590 570mg | TLC590 475mg | Naropin 150mg
Started | 12 | 0 | 0 | 0 | 4
Completed | 12 | 0 | 0 | 0 | 3
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1
Period: TLC590 380mg and Naropin 150mg
Arm/Group | TLC590 190mg | TLC590 380mg | TLC590 570mg | TLC590 475mg | Naropin 150mg
Started | 0 | 12 | 0 | 0 | 5
Completed | 0 | 11 | 0 | 0 | 4
Not Completed | 0 | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1
Period: TLC590 570mg and Naropin 150mg
Arm/Group | TLC590 190mg | TLC590 380mg | TLC590 570mg | TLC590 475mg | Naropin 150mg
Started | 0 | 0 | 12 | 0 | 4
Completed | 0 | 0 | 11 | 0 | 3
Not Completed | 0 | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 1
Period: TLC590 475mg and Naropin 150mg
Arm/Group | TLC590 190mg | TLC590 380mg | TLC590 570mg | TLC590 475mg | Naropin 150mg
Started | 0 | 0 | 0 | 12 | 4
Completed | 0 | 0 | 0 | 12 | 4
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: One subject who was randomized (period 2, Naropin group) did not receive any treatment (withdraw by subject), and was replaced. This subject was not included in any analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | TLC590 190mg | TLC590 380mg | TLC590 570mg | TLC590 475mg | Naropin 150mg | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 16 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 12 | 12 | 16 | 64
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 2 | 1 | 4
  Male | 12 | 11 | 12 | 10 | 15 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 12 | 12 | 12 | 16 | 63
  Not Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 12 | 12 | 12 | 16 | 64
Body Mass Index (BMI) [Count of Participants; unit: Participants]
  BMI <=35 kg/m2 | 12 | 12 | 12 | 12 | 16 | 64
  BMI > 35 kg/m2 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability: Event of SAE and Treatment-related Severe AE
Description: Event of serious adverse event (SAE) and treatment-related severe adverse event (TRAE)
Time Frame: Screening till 30 days post investigational product (IP) administration, up to 58 days
Measure: Number; unit: Event
Groups:
- TLC570mg; TLC590 475mg: TLC590 (Ropivacaine Liposome Injectable Suspension) is a sustained-release liposome formulation of ropivacaine, white aqueous suspension with ropivacaine concentration at approximately 19 mg/mL.
  TLC590: TLC590 lyophilized cake will be reconstituted with the TLC590 reconstitution solution to form the TLC590 ropivacaine liposome injectable suspension
- Naropin: Naropin injection contains ropivacaine HCl. Strength: 150mg/ 30mL (5 mg/mL) Size: 30mL fill, in a 30mL single dose vial
  Naropin: Local infiltration of Naropin to produce anesthesia for surgery and analgesia in postoperative pain management. Naropin 150mg [0.5%, 5mg/mL] x 30mL
Arm/Group | TLC590 190mg | TLC590 380mg | TLC570mg | TLC590 475mg | Naropin
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 16
Event | 2 | 1 | 2 | 2 | 2

ADVERSE EVENTS:
Time Frame: 58 days
Description: Total 64 subjects were enrolled in the study, 12 subjects in each TLC590 group and 16 subjects in Naropin group.
Groups:
- TL590 570mg; TLC590 475mg: TLC590 (Ropivacaine Liposome Injectable Suspension) is a sustained-release liposome formulation of ropivacaine, white aqueous suspension with ropivacaine concentration at approximately 19 mg/mL.
  TLC590: TLC590 lyophilized cake will be reconstituted with the TLC590 reconstitution solution to form the TLC590 ropivacaine liposome injectable suspension
Arm/Group | TLC590 190mg | TLC590 380mg | TL590 570mg | TLC590 475mg | Naropin 150mg
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/16
Other Adverse Events (participants affected / at risk) | 11/12 | 8/12 | 7/12 | 10/12 | 13/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TLC590 190mg (N=12) | TLC590 380mg (N=12) | TL590 570mg (N=12) | TLC590 475mg (N=12) | Naropin 150mg (N=16)
Nausea (Gastrointestinal disorders) | 4 (5) | 2 (3) | 2 (3) | 5 (5) | 7 (7)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 8 (8)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (3) | 0 (0) | 2 (2) | 5 (5)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 4 (4) | 3 (3)
Dizziness (Nervous system disorders) | 2 (4) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incision site hypoaesthesia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural dizziness (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pallor (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epididymitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QRS complex prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Electrocardiogram ST-T change (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram T wave inversion (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Testicular oedema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Unless Sponsor provides prior written consent, Institution may not use Confidential Information for any purpose other than that authorized in this Agreement, nor may Institution disclose Confidential Information to any third party except as authorized in this Agreement or as required by law. Required disclosure of Confidential Information to the Institutional Review Board (IRB) or to FDA representatives is specifically authorized.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-13): https://cdn.clinicaltrials.gov/large-docs/46/NCT03591146/Prot_SAP_000.pdf